CLINICAL TRIAL: NCT04468672
Title: The Interaction of Shift Work and Food Environment on Eating Behaviors and Appetite
Brief Title: Eating Behaviors in Shift Workers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor of Nutritional Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS8559
Record Dates: First submitted 2020-06-30; First posted 2020-07-13 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Shift Work Type Circadian Rhythm Sleep Disorder; Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Portion Size

STUDY DESIGN:
Intervention Model Description: This is a mixed design with two participant groups (between-subject), day and night workers, each being exposed to 4 levels of food portion size (within-subjects factor)
Who Masked: Outcomes Assessor
Masking Description: Statistician will be blinded to participant group and condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day worker (Active Comparator): Men and women who work only day shift for at least 3 consecutive days of the week
  Interventions: Behavioral: Portion size
- Night worker (Active Comparator): Men and women who work only night shift for at least 3 consecutive days of the week
  Interventions: Behavioral: Portion size

INTERVENTIONS:
Behavioral: Portion size — The amount of food served (g) at the first two meals of each day. These amounts will vary across 4 weeks.

SUMMARY:
This study will compare eating behaviors and measures of hunger and fullness between day and night workers in order to better understand why night workers are at increased risk for obesity and related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Work ~ 8-hour shifts during day or night on 3 or more consecutive days of the week
* BMI 19-35 kg/m^2
* Age 20-55 years of age
* Metabolically healthy
* Weight stable over previous 3 months
* Lives in New York City area

Exclusion Criteria:

* Pregnant or less than 1 year postpartum at time of study
* Smoking
* History of drug or alcohol abuse
* Rotating shift work
* Habitual sleep duration of more than 6 hour per night
* Obstructive sleep apnea
* Transmeridian travel
* Type 2 diabetes
* Cardiovascular disease
* Hypertension
* Participation in diet or weight loss program in the 3 months prior to enrollment
* Psychiatric or sleep disorder
* Food allergies or intolerances
* Dislike of or unwillingness to eat test foods

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Food intake | 24-hours intake period
  Food by weight (g) in response to variations in portion served
Energy intake | 24-hours intake period
  Food by energy (kcal) in response to variations in portion served
Energy density consumed | 24-hours intake period
  Energy density consumed (kcal/g) in response to variations in portion served

SECONDARY OUTCOMES:
Appetite-regulating hormones | 2-hours measurement period
  Appetite-regulating hormones, including Glucagon-like-peptide 1 (GLP-1) and ghrelin will be analyzed from plasma from whole blood samples collected while fasted and at 30, 60, 90, and 120 min postprandial. Area under the curve of plasma concentrations will be calculated for each individual appetite-regulating hormone
Hunger and fullness | 24-hours measurement period
  Subjective measures related to hunger, fullness, and prospective consumption will be measured before and after meals via visual analog scales. The range of scores are 0 mm to 100 mm, with higher scores indicating greater feelings of the corresponding measure (e.g. greater hunger). Post-meal measures, adjusted for the corresponding pre-meal measure, will be analyzed as individual outcomes. Area under the curve will also be calculated for each measure.

CONTACTS AND LOCATIONS:
Overall Officials: Faris M Zuraikat, PhD, Principal Investigator — Columbia University; Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study is completed (data collection, analysis, publication) and after any subsequent funding applications have been submitted.
Access Criteria: Upon request